CLINICAL TRIAL: NCT02248311
Title: "Preventing Cardiovascular Ischemic Events and Arresting Their Consequences in Type 2 Diabetic Population: a Multidisciplinary Clinical and Experimental Approach" (PRECISED)
Brief Title: "Preventing Cardiovascular Ischemic Events and Arresting Their Consequences in Type 2 Diabetic Population
Acronym: PRECISED
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PRECISED ISCiii-PIE-13
Record Dates: First submitted 2014-09-18; First posted 2014-09-25 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Type2 Diabetes Mellitus; Microangiopathy; Non Alcoholic Fatty Liver Disease; Coronary Artery Disease; Cerebrovascular Disease; Acute Coronary Syndrome/ Myocardial Infarction; Ictus
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Coronary Artery Disease; Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Patients: 200 Control group: 60
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients/Control Group: Observational
- Patients/Group Control: Observational

SUMMARY:
Current methods based on traditional Cardiovascular risk factors are not clinically useful for identifying Type 2 Diabetes patients at risk of developing acute Cardiovascular ischemic events (ie.myocardial infarction or stroke). In addition, Cardiovascular ischemic events in Type 2 Diabetes population have worse prognosis than in general population. In fact, there is sufficient experimental evidence indicating that diabetes exaggerates the deleterious effects of ischemic events and worsens their outcome.

A prolonged sub-clinical phase exists before a Cardiovascular event occurs in Type 2 Diabetes patients. Therefore, new strategies aimed at identifying those patients with this subclinical Cardiovascular Diabetes and, consequently, more prone to develop Cardiovascular events is a challenge to be met.

DETAILED DESCRIPTION:
Objectives

1) To examine whether the extension and degree of microangiopathy is an independent risk factor for silent myocardial and brain ischemia. 2) To evaluate whether the degree and extension of microangiopathy is a predictor of CV events and poor outcome. 3) To evaluate whether a new score based on the extension and the degree of microangiopathy will permit us to improve the current methods used to identify patients at risk of CVD and its outcomes. 4) To determine whether the presence and the degree of NAFLD is an independent Cardiovascular disease risk factor and represent and extra-value to the score based on the extension and the degree of microangiopathy.

Secondary objectives:

1) To examine the usefulness of selected serum biomarkers in identifying diabetic patients at risk of Cardiovascular disease 2) To evaluate whether these selected biomarkers are related to the degree and extension of microangiopathy and the outcome of cardiovascular events. 3) To better define the meaning of microalbuminuria in type 2 diabetic population (glomerular involvement vs. index of generalized endothelial dysfunction)

ELIGIBILITY:
Inclusion Criteria:

* a) Age from 50-79 years; b) History of type 2diabetes of at least one year. Diabetes will be defined following the American Diabetic Association criteria: fasting glucose level of at least 126 mg/dl [7.0 mmol/l] in two separate analyses, a non-fasting glucose level of at least 200 mg/dl [11.1 mmol/l] or a self-reported history of physician-diagnosed diabetes or treatment for diabetes

Exclusion Criteria:

* a) Past medical history of Cardiovascular event; b) Type 1 diabetes; c) Contraindication for PET-CT or MRI d) Other concomitant disease associated with a short life expectancy

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 200 T2D diabetic patients without history of clinical Cardiovascular disease will be recruited from the Outpatient Diabetic Clinic of Vall d'Hebron Hospital and the Primary Health Care centers under its influence area. Sixty non-diabetic patients without classic Cardiovascular risk factors matched by age will be used as a control group. Specifically, vascular risk factors, concomitant diseases, family history of Cardiovascular disease or stroke and the treatments taken at the time of inclusion will be collected.
Sampling Method: Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2014-09; Primary Completion 2018-02 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Subclinical Cardiovascular Diseases | 1 week
  Number of Type 2 Diabetes (T2D) patients presenting subclinical Cardiovascular disease as defined by the presence of brain infarcts (MRI), myocardial infarcts, or myocardial ischemia or > 50% coronary artery stenosis (PET-SPECT)

SECONDARY OUTCOMES:
Ischemic events | 3 years
  * Occurrence of Cardiovascular events during the 3 year follow up: Ictus, transient ischemic attack, acute coronary syndrome (STEMI or NSTEMI), angina, sudden cardiac death.
  * Incidence of major adverse cardiovascular events at 30 days following acute ischemic syndrome (Death, Re-infarction, Ictus)

CONTACTS AND LOCATIONS:
Overall Officials: David García-Dorado Garcia, PhD MD, Principal Investigator — Hospital Universitario Valle de Hebron, Barcelona, Spain; Joan Montaner Vilallonga, PhD MD, Principal Investigator — Hospital Universitario Valle de Hebron, Barcelona, Spain; Rafael Simó Canonge, PhD MD, Principal Investigator — Hospital Universitario Valle de Hebron, Barcelona, Spain; Joan Sayós Ortega, PhD MD, Principal Investigator — Hospital Universitario Valle de Hebron, Barcelona, Spain; Daniel Serón Micas, PhD MD, Principal Investigator — Hospital Universitario Valle de Hebron, Barcelona, Spain; Joan Genescà Ferrer, PhD MD, Principal Investigator — Hospital Universitario Valle de Hebron, Barcelona, Spain; Santiago Aguadé Bruix, PhD MD, Principal Investigator — Hospital Universitario Valle de Hebron, Barcelona, Spain; Joan Xavier Comella Carnicé, PhD MD, Principal Investigator — Hospital Universitario Valle de Hebron, Barcelona, Spain
Locations (1):
- Hospital Universitario Valle de Hebron, Barcelona, Spain